CLINICAL TRIAL: NCT02034799
Title: A Prospective, Randomized, Controlled Phase IV Study to Compare Bioseal Versus Standard of Care as an Adjunct to Hemostasis in Elective Brain Tumor Surgery
Brief Title: Phase IV Bioseal Study in Brain Tumor Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ethicon, Inc. (Industry)
Collaborators: Guangzhou Bioseal Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BIOS-13-002
Record Dates: First submitted 2014-01-10; First posted 2014-01-14 (Estimated); Results first posted 2018-02-26 (Actual); Last update posted 2018-02-26 (Actual); Status verified 2017-08

CONDITIONS: Hemostasis; Meningioma Surgery
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (SoC) (Other): Standard of Care (SoC) include any active or inactive adjunctive treatment to hemostasis methods currently used based on each surgeons surgical practice except for the use of other fibrin sealants.
  Interventions: Other: Standard of Care (SoC)
- Bioseal Fibrin Sealant (Experimental): A porcine-derived fibrin sealant consisting of thrombin and fibrinogen
  Interventions: Biological: Bioseal Fibrin Sealant

INTERVENTIONS:
Biological: Bioseal Fibrin Sealant
  Arms: Bioseal Fibrin Sealant
Other: Standard of Care (SoC)
  Arms: Standard of Care (SoC)

SUMMARY:
The objective of this study is to observe the clinical utility and performance of Bioseal when used as an adjunct to hemostasis versus Standard of Care (SoC) in elective meningioma surgery.

ELIGIBILITY:
Inclusion Criteria:

* Subjects between 18 and 75 years of age
* Undergoing elective meningioma surgery and having a tumor cavity
* Presence of an appropriate Target Bleeding Site (TBS) as identified intra-operatively by the surgeon requiring an adjunct to achieve hemostasis
* Able and willing to comply with procedures required by protocol
* Signed and dated written informed consent prior to any study related procedures.

Exclusion Criteria:

* Subjects undergoing emergency surgery
* Subjects with any intra-operative findings that may preclude conducting of the study procedures
* Intended use of Fibrin Sealants (including autologous Fibrin Sealants) other than Bioseal on the Target Bleeding Site (TBS)
* Subjects with known intolerance to blood products or to one of the components of the study product or unwilling to receive blood products
* Subjects who have a history of traumatic head injury
* Female subjects who are known breastfeeding or pregnant or intend to become pregnant during the clinical study period
* The subject, in the opinion of the investigator, would not be suitable for participation in the study
* Subjects who participated in another trial within 30 days prior to the planned start of treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2013-11-01 (Actual); Primary Completion 2014-08-01 (Actual); Study Completion 2014-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Kocharian, MD, PhD, Study Director — Ethicon, Inc.
Locations (7):
- China (7):
  - Clinical Investigation Site #6, Zhengzhou, Henan
  - Clinical Investigation Site #5, Changsha, Hunan
  - Clinical Investigation Site #3, Chengdu, Sichuan
  - Clinical Investigation Site #4, Hangzhou, Zhejiang
  - Clinical Investigation Site #7, Beijing
  - Clinical Investigation Site #2, Shanghai
  - Clinical Investigation Site #1, Tianjin

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard of Care (SoC): SoC include Standard of Care (SoC) included manual compression, cautery, manual compression and cautery with a non-fibrin sealant topical absorbable hemostat (TAH).
Period: Overall Study
Arm/Group | Standard of Care (SoC) | Bioseal Fibrin Sealant
Started | 129 | 127
Completed | 127 | 123
Not Completed | 2 | 4
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Death | 2 | 1

BASELINE CHARACTERISTICS:
Population: Adult subjects between the ages of 18 and 75 years were eligible for recruitment into the study.Subject 16225 was enrolled at age 12 and did not match the study inclusion/exclusion criteria. This was logged as a protocol deviation.
Groups:
- Standard of Care (SoC): Standard of Care (SoC) included manual compression, cautery, manual compression and cautery with a non-fibrin sealant topical absorbable hemostat (TAH). Standard of Care (SoC)
- Bioseal Fibrin Sealant: A porcine-derived fibrin sealant consisting of thrombin and fibrinogen Bioseal Fibrin Sealant
- Total: Total of all reporting groups
Arm/Group | Standard of Care (SoC) | Bioseal Fibrin Sealant | Total
Number analyzed (Participants) | 129 | 127 | 256
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 1
  Between 18 and 65 years | 106 | 98 | 204
  >=65 years | 23 | 28 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.9 (11.3) | 50.7 (11.7) | 49.8 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 80 | 149
  Male | 60 | 47 | 107
Height [Mean (Standard Deviation); unit: cm] | 164.5 (7.0) | 163.6 (7.6) | 164.1 (7.3)
Height [Median (Full Range); unit: cm] | 163 [152 to 180] | 161 [141 to 180] | 162 [141 to 180]
Weight [Mean (Standard Deviation); unit: kg] | 62.9 (10.3) | 62.2 (8.8) | 62.6 (9.6)
Weight [Median (Full Range); unit: kg] | 62 [45 to 98] | 60 [40 to 85] | 61 [40 to 98]
BMI [Mean (Standard Deviation); unit: (kg/m^2)] | 23.2 (3.4) | 23.2 (2.8) | 23.2 (3.1)
BMI [Median (Full Range); unit: (kg/m^2)] | 22.5 [17.8 to 34.7] | 23.1 [17.0 to 31.2] | 22.8 [17.0 to 34.7]
BMI Group [Number; unit: participants]
  Underweight | 3 | 2 | 5
  Normal | 96 | 95 | 191
  Overweight | 22 | 27 | 49
  Obese | 8 | 3 | 11
Smoking Status [Number; unit: participants]
  Current Smoker | 18 | 12 | 30
  Former Smoker | 4 | 3 | 7
  Never Smoked | 107 | 112 | 219

OUTCOME MEASURES:

1. Primary Outcome: Hemostasis at the Target Bleeding Site (TBS) at 6 Minutes Following Treatment Application. Hemostasis is Defined as no Detectable Bleeding at the TBS.
Description: The percentage of participants with hemostasis at the Target Bleeding Site (TBS) at 6 minutes following start of treatment application. Hemostasis is defined as no detectable bleeding at the TBS.
Time Frame: Intra-operative, 6 minutes following randomization
Measure: Number (95% Confidence Interval); unit: % of participants
Groups:
- Standard of Care (SoC): Standard of Care (SoC) included manual compression, cautery, manual compression and cautery with a non-fibrin sealant topical absorbable hemostat (TAH).
Arm/Group | Standard of Care (SoC) | Bioseal Fibrin Sealant
Number analyzed (Participants) | 129 | 127
% of participants | 99.2 [95.8 to 100] | 100 [97.1 to 100]
Statistical Analysis 1: Comparison: Standard of Care (SoC) vs Bioseal Fibrin Sealant; H0: Delta </= -0.1 HA: Delta > -0.1 Delta is difference in proportion of successes between Bioseal and SOC gropus (Bioseal minus SOC). Success is defined as hemostasis at the TBS at 6 minutes following treatment application; Test type: Non-Inferiority or Equivalence — The assumed proportion of success for SOC is 0.95 and the proportion of success for the Bioseal group at which the power is calculated is 0.95. A sample size of 112 subjects per group achieves 80% power to detect the non-inferiority margin difference between the group proportions of -0.10. One-sided significance level of 0.025 was used. Using drop-out rate of 10%, 125 subjects per treatment group were randomized for a total of 250 subjects; Risk Difference (RD) = 0.0781, 95% CI 2-sided [-0.048 to 0.199]

2. Secondary Outcome: Hemostasis at the TBS at 3 Minutes Following Treatment Application
Description: The percentage of participants with hemostasis at the Target Bleeding Site (TBS) at 3 minutes following start of treatment application. Hemostasis was defined as no detectable bleeding at the TBS.
Time Frame: Intra-operative, 3 minutes following randomization
Measure: Number (95% Confidence Interval); unit: % of participants
Arm/Group | Standard of Care (SoC) | Bioseal Fibrin Sealant
Number analyzed (Participants) | 129 | 127
% of participants | 89.9 [83.4 to 94.5] | 94.5 [89.0 to 97.8]

3. Secondary Outcome: Incidence of Neurosurgical Complications, Central Nervous System Events and Surgical Wound Complications.
Time Frame: Through 30-day follow-up
Measure: Number; unit: participants
Arm/Group | Standard of Care (SoC) | Bioseal Fibrin Sealant
Number analyzed (Participants) | 129 | 127
participants
  Neurosurgical Complication | 14 | 14
  Unplanned Intervention | 5 | 3
  Central Nervous System | 6 | 8
  Surgical Wound Complication | 5 | 3

4. Secondary Outcome: Incidence of Potential Bleeding-related Adverse Events
Time Frame: Through 30-day follow-up
Measure: Number; unit: participants
Arm/Group | Standard of Care (SoC) | Bioseal Fibrin Sealant
Number analyzed (Participants) | 129 | 127
participants | 18 | 18

ADVERSE EVENTS:
Time Frame: Adverse events were assessed and recorded from the time of treatment application until completion of the 30 (± 7) days follow up period.
Arm/Group | Standard of Care (SoC) | Bioseal Fibrin Sealant
Serious Adverse Events (participants affected / at risk) | 10/129 | 5/127
Other Adverse Events (participants affected / at risk) | 22/129 | 26/127
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care (SoC) (N=129) | Bioseal Fibrin Sealant (N=127)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Postoperative Wound Infection (Infections and infestations) | 1 (1) | 1 (1)
Brain Herniation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Extradural Haematoma (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Head Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural Haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fibrinolysis (Investigations) | 1 (1) | 0 (0)
Glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant Neoplasm Progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Brain Oedema (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral Ischaemia (Nervous system disorders) | 1 (1) | 1 (1)
VIIth Nerve Paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care (SoC) (N=129) | Bioseal Fibrin Sealant (N=127)
Anemia (Blood and lymphatic system disorders) | 8 (8) | 11 (11)
Pyrexia (General disorders) | 4 (4) | 7 (7)
Lung Infection (Infections and infestations) | 7 (7) | 2 (2)
Brain Oedema (Nervous system disorders) | 8 (8) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less